CLINICAL TRIAL: NCT00111410
Title: A Multicenter, Double-Blind, Randomized, Placebo Controlled Study to Estimate the Effect of Anakinra (r-metHuIL-1ra) on Vaccine Antibody Response in Subjects With Rheumatoid Arthritis (RA)
Brief Title: Evaluating the Effect of Anakinra (r-metHuIL-1ra) on Vaccine AntibodyResponse in Subjects With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Organization: Swedish Orphan Biovitrum (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20020101
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Inflammation; Interleukin-1 (IL-1), r-metHuIL-1ra; Autoimmune, Kineret®; Anakinra, Immunex; Amgen, Clinical Trials
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

INTERVENTIONS:
Drug: Anakinra (r-metHuIL-1ra)

SUMMARY:
The purpose of this study is to estimate the effect of anakinra, 100 mg once daily (QD), on the development of an anti-tetanus antibody response in subjects with RA after vaccination with a tetanus and diphtheria toxoids injection. In addition, this study will evaluate the general safety profile of therapy with anakinra, 100 mg QD, in subjects with RA after vaccination with a tetanus and diphtheria toxoids injection.

ELIGIBILITY:
Inclusion Criteria: - Diagnosed with RA by American College of Rheumatology (ACR) criteria for greater than or equal to 12 weeks - Active RA with at least 3 swollen joints and 3 tender/painful joints and at least one of the following:

* Morning stiffness greater than or equal to 45 minutes;
* C-reactive protein (CRP) greater than or equal to 1.5 mg/dL;
* Erythrocyte sedimentation rate greater than or equal to 28 mm/hr;
* Stable methotrexate dose of less than or equal to 20 mg/week for 8 weeks prior to randomization;
* Stable doses of nonsteroidal anti-inflammatory drugs (NSAIDs) and oral corticosteroids (less than or equal to 10 mg/day of prednisone or equivalent) for 4 weeks prior to randomization. Exclusion Criteria: - Pregnant or breast-feeding women - Any uncontrolled, clinically significant systemic disease - Has total white cell count less than 3.5 x 10^9/L, a neutrophils count less than 2.0 x 10^9/L, platelet count less than 125 x 10^9/L or hemoglobin (Hgb) less than 8.0 g/dL at screening - Abnormal liver function tests (AST/ALT greater than or equal to 1.5 x the upper limit of normal at screening) - Serum creatinine greater than 1.5 x the upper limit of normal at screening - Subject recall of having tetanus toxoid or diphtheria vaccination less than 10 years prior to randomization - Has never received a primary tetanus vaccination - Any other vaccination within 12 weeks of randomization - Disease-modifying antirheumatic drugs (DMARDs) other than methotrexate - Biologics to treat RA within the previous 8 weeks of screening (e.g., etanercept, infliximab) - Subjects were treated with anakinra within 4 weeks prior to randomization

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects that achieve an anti-tetanus antibody response rate at study week 8 (4 weeks after the tetanus injection), based on a 4-fold titer development relative to week 4 (pre-vaccination)

SECONDARY OUTCOMES:
Anti-tetanus antibody titers at weeks 4 and 8
Anti-tetanus antibody level changes from baseline to week 4
Anti-tetanus antibody level changes from week 4 to week 8
Antibody level of at least 0.1 IU/mL at week 8.
Safety evaluation of serious adverse events, adverse events and laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com